CLINICAL TRIAL: NCT00501046
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of AST-120 for Prevention of Chronic Kidney Disease Progression in Patients With Moderate to Severe Chronic Kidney Disease Including Assessment of Quality of Life
Brief Title: A Study of AST-120 for Evaluating Prevention of Progression In Chronic Kidney Disease Including Assessment of Quality of Life (EPPIC-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Kureha Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRM-307
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — AST 120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AST-120 (Experimental)
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: Placebo — 9g /day (3 times a day)
  Arms: Placebo
Drug: AST-120 — 9g /day (3 times a day)
  Arms: AST-120

SUMMARY:
1) To evaluate the effectiveness of AST-120 (spherical carbon adsorbent) added to standard-of-care therapy in moderate to severe Chronic Kidney Disease (CKD), on time to first occurrence of any event of the triple composite outcome of initiation of dialysis, kidney transplant or doubling of serum creatinine (sCr) when compared with placebo; 2) To evaluate the safety and tolerability of long-term AST-120 therapy in patients with CKD; 3) To evaluate the effects of AST-120 versus placebo, on other measures of renal function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Moderate to severe CKD, not anticipated to require dialysis or renal transplant within the next 6 months
* Patient survival expected to be no less than one year
* Serum creatinine in men >= 2.0 mg/dL (>= 177 µmol/L) and <= 5.0 mg/dL (<= 442 µmol/L), and in women >= 1.5 mg/dL (>= 133 µmol/L) and <= 5.0 mg/dL (<= 442 µmol/L) at Screening
* Urinary total protein to urinary total creatinine ratio must be >= 0.5 on a spot void obtained at Screening
* Blood pressure <= 160/90 mmHg at both Screening and Baseline visits. In addition, blood pressure, if measured, must have been stable in hypertensive patients over the 3 months prior to Screening, with no more than 1 blood pressure reading > 160/90 mmHg
* In patients being treated for hypertension, they should be on a stable anti-hypertensive regimen

Exclusion Criteria:

* Obstructive or reversible cause of kidney disease
* Nephrotic syndrome defined as a ratio of urinary total protein to urinary creatinine of > 6.0 as measured on a spot void
* Adult polycystic kidney disease
* History of previous kidney transplant
* History of recent (within the past 6 months) accelerated or malignant hypertension
* Uncontrolled arrhythmia or severe cardiac disease within the past 6 months
* History of malabsorption, inflammatory bowel disease, hiatal hernia, active peptic ulcer, or severe GI dysmotility, not attributable to the use of a phosphate binder
* Received any investigational agent or participated in a clinical study within the previous 3 months
* Presence of any significant medical condition that might create an undue risk with study participation, or significantly confound the collection of safety and efficacy data in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2007-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Tanabe Pharma Development America, Inc.
Locations (106):
- United States (46):
  - Tuscaloosa, Alabama
  - Hot Springs, Arkansas
  - Bakersfield, California
  - Glendale, California
  - Los Angeles, California
  - Palo Alto, California
  - Riverside, California
  - Denver, Colorado
  - Boynton Beach, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Macon, Georgia
  - Honolulu, Hawaii
  - Evergreen Park, Illinois
  - Shawnee Mission, Kansas
  - Kenner, Louisiana
  - Shreveport, Louisiana
  - Pontiac, Michigan
  - Brooklyn Center, Minnesota
  - Flushing, New York
  - Great Neck, New York
  - New York, New York
  - Williamsville, New York
  - Elizabeth City, North Carolina
  - Cincinnati, Ohio
  - Bend, Oregon
  - Allentown, Pennsylvania
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Arlington, Virginia
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Vancouver, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - San Miguel de Tucumán
- Brazil (9):
  - Belo Horizonte
  - Botucatu
  - Campinas
  - Curitiba
  - Ibirapuera
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
  - Sorocaba
- Canada (4):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Greenfield Park, Quebec
  - Montreal, Quebec
- Czechia (4):
  - Hradec Králové
  - Liberec
  - Prague
  - Ústí nad Labem
- Germany (3):
  - Hamburg
  - Kiel
  - Mainz
- Mexico (5):
  - Aguascalientes
  - Cuernavaca
  - Durango
  - Mexico City
  - México
- Poland (4):
  - Bialystok
  - Częstochowa
  - Lublin
  - Warsaw
- San Juan, Puerto Rico
- Russia (12):
  - Arkhangelsk
  - Chelyabinsk
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Orenburg
  - Petrozavodsk
  - Saint Petersburg
  - Saratov
  - Tomsk
  - Yaroslayl
  - Yekaterinburg
- Spain (5):
  - A Coruña
  - Asturias
  - Barcelona
  - Guadalajara
  - Madrid
- Ukraine (10):
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Luhansk
  - Lviv
  - Mykolayiv
  - Poltava
  - Ternopil
  - Vinnitsa
  - Zaporizhzhya

REFERENCES:
- [Result] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Arita K, Kato A, Shimizu M. Randomized Placebo-Controlled EPPIC Trials of AST-120 in CKD. J Am Soc Nephrol. 2015 Jul;26(7):1732-46. doi: 10.1681/ASN.2014010042. Epub 2014 Oct 27. PMID 25349205
- [Derived] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Shimizu M, Kikuchi M, Shobu Y. Risk factors for progression of chronic kidney disease in the EPPIC trials and the effect of AST-120. Clin Exp Nephrol. 2018 Apr;22(2):299-308. doi: 10.1007/s10157-017-1447-0. Epub 2017 Jul 24. PMID 28741050
- [Derived] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Shimizu M, Shobu Y, Kikuchi M. The effects of AST-120 on chronic kidney disease progression in the United States of America: a post hoc subgroup analysis of randomized controlled trials. BMC Nephrol. 2016 Sep 30;17(1):141. doi: 10.1186/s12882-016-0357-9. PMID 27716149

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AST-120 | Placebo
Started | 508 | 507
Completed | 238 | 213
Not Completed | 270 | 294
Not completed — Adverse Event | 21 | 25
Not completed — Death | 23 | 30
Not completed — Lost to Follow-up | 14 | 13
Not completed — Physician Decision | 7 | 2
Not completed — Pregnancy | 0 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 84 | 83
Not completed — Reaching endpoints,Noncompliance,etc | 119 | 137

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AST-120 | Placebo | Total
Number analyzed (Participants) | 508 | 507 | 1015
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (15.52) | 55.7 (14.66) | 55.1 (15.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 226 | 455
  Male | 279 | 281 | 560

OUTCOME MEASURES:

1. Primary Outcome: Composite of Dialysis Initiation, Kidney Transplantation, and Serum Creatinine Doubling. Number of Participants Meeting the Criteria Are Reported.
Time Frame: Beyond Week 48, a 12-week visit cycle continued until the end of the study or until individual patients reached an endpoint
Population: ITT (censored at last contact)
Measure: Number; unit: participants
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 500 | 497
participants | 172 | 183

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events and Treatment-emergent Serious Adverse Events
Time Frame: Approximately 42 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
Participants
  Treatment-emergent AE | 438 | 425
  Treatment-emergent SAE | 156 | 178

3. Secondary Outcome: Number of Participants Who Developed a Component of a Quadruple Composite Endpoint (Initiation of Dialysis, Kidney Transplant, Doubling of sCr, or Death)
Time Frame: approximately 42 months
Population: ITT (censored at last contact)
Measure: Count of Participants; unit: Participants
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 500 | 497
Participants | 204 | 217

4. Secondary Outcome: Vitamin A Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 430.293 Days), Final Visit (Mean: 908.486 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
ng/mL
  Baseline: number analyzed (Participants) | 469 | 453
  Baseline | 1143.6 (398.42) | 1159.4 (404.85)
  Week 12: number analyzed (Participants) | 439 | 430
  Week 12 | 1098.9 (376.33) | 1182.9 (411.38)
  Week 24: number analyzed (Participants) | 427 | 410
  Week 24 | 1106.0 (371.04) | 1180.5 (385.83)
  Week 36: number analyzed (Participants) | 409 | 396
  Week 36 | 1118.4 (382.22) | 1201.6 (401.03)
  Week 48: number analyzed (Participants) | 385 | 371
  Week 48 | 1117.0 (380.72) | 1196.7 (399.97)
  Week 60: number analyzed (Participants) | 362 | 332
  Week 60 | 1162.6 (373.49) | 1242.3 (421.19)
  Week 72: number analyzed (Participants) | 335 | 303
  Week 72 | 1157.6 (397.82) | 1243.5 (416.84)
  Week 84: number analyzed (Participants) | 305 | 274
  Week 84 | 1225.6 (418.23) | 1249.3 (379.41)
  Week 96: number analyzed (Participants) | 236 | 207
  Week 96 | 1219.5 (419.49) | 1267.8 (376.38)
  Week 108: number analyzed (Participants) | 190 | 166
  Week 108 | 1231.2 (397.68) | 1266.6 (427.25)
  Week 120: number analyzed (Participants) | 146 | 132
  Week 120 | 1240.8 (387.79) | 1198.7 (388.77)
  Week 132: number analyzed (Participants) | 114 | 91
  Week 132 | 1253.2 (376.03) | 1234.2 (365.55)
  Week 144: number analyzed (Participants) | 78 | 70
  Week 144 | 1324.6 (567.01) | 1204.5 (414.34)
  Week 156: number analyzed (Participants) | 51 | 48
  Week 156 | 1196.3 (456.16) | 1193.0 (389.27)
  Week 168: number analyzed (Participants) | 35 | 24
  Week 168 | 1265.0 (478.26) | 1363.7 (348.93)
  Week 180: number analyzed (Participants) | 15 | 13
  Week 180 | 1243.4 (454.73) | 1147.8 (254.30)
  Early Term/ Discontinuation: number analyzed (Participants) | 97 | 111
  Early Term/ Discontinuation | 1231.2 (442.79) | 1269.4 (425.09)
  Final Visit: number analyzed (Participants) | 229 | 207
  Final Visit | 1223.3 (393.07) | 1274.5 (350.67)

5. Secondary Outcome: Vitamin B12 Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 425.112 Days), Final Visit (Mean: 910.988 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
pg/mL
  Baseline: number analyzed (Participants) | 498 | 490
  Baseline | 651.7 (1961.13) | 747.9 (2521.02)
  Week 12: number analyzed (Participants) | 462 | 448
  Week 12 | 497.6 (1466.88) | 464.3 (650.01)
  Week 24: number analyzed (Participants) | 436 | 415
  Week 24 | 608.4 (2016.76) | 681.0 (2127.01)
  Week 36: number analyzed (Participants) | 410 | 393
  Week 36 | 631.8 (2079.77) | 618.7 (2031.35)
  Week 48: number analyzed (Participants) | 385 | 367
  Week 48 | 455.2 (371.17) | 728.4 (2412.07)
  Week 60: number analyzed (Participants) | 357 | 330
  Week 60 | 444.4 (332.65) | 637.8 (1911.72)
  Week 72: number analyzed (Participants) | 334 | 293
  Week 72 | 601.6 (1882.39) | 741.3 (2281.81)
  Week 84: number analyzed (Participants) | 305 | 272
  Week 84 | 465.2 (637.01) | 740.9 (2492.87)
  Week 96: number analyzed (Participants) | 235 | 208
  Week 96 | 444.8 (364.90) | 459.5 (548.84)
  Week 108: number analyzed (Participants) | 189 | 166
  Week 108 | 700.2 (2110.74) | 505.6 (771.70)
  Week 120: number analyzed (Participants) | 148 | 132
  Week 120 | 509.9 (726.72) | 689.1 (1864.40)
  Week 132: number analyzed (Participants) | 113 | 90
  Week 132 | 657.7 (1428.09) | 476.9 (483.88)
  Week 144: number analyzed (Participants) | 77 | 70
  Week 144 | 416.3 (211.52) | 721.3 (1543.37)
  Week 156: number analyzed (Participants) | 51 | 47
  Week 156 | 601.5 (744.06) | 1046.6 (3595.42)
  Week 168: number analyzed (Participants) | 35 | 24
  Week 168 | 552.7 (570.85) | 750.2 (1385.54)
  Week 180: number analyzed (Participants) | 15 | 13
  Week 180 | 494.5 (389.57) | 1062.7 (2386.40)
  Early Term/ Discontinuation: number analyzed (Participants) | 95 | 111
  Early Term/ Discontinuation | 1186.2 (4148.50) | 1174.8 (3403.80)
  Final Visit: number analyzed (Participants) | 228 | 205
  Final Visit | 764.2 (2392.88) | 505.5 (1063.91)

6. Secondary Outcome: 25-Hydroxyvitamin D Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 429.695 Days), Final Visit (Mean: 908.601 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
ng/mL
  Baseline: number analyzed (Participants) | 503 | 502
  Baseline | 21.09 (10.391) | 20.36 (10.063)
  Week 12: number analyzed (Participants) | 474 | 463
  Week 12 | 21.64 (9.981) | 21.08 (10.246)
  Week 24: number analyzed (Participants) | 446 | 427
  Week 24 | 21.70 (10.166) | 21.28 (10.100)
  Week 36: number analyzed (Participants) | 415 | 398
  Week 36 | 21.72 (10.441) | 21.00 (9.766)
  Week 48: number analyzed (Participants) | 391 | 369
  Week 48 | 21.10 (10.195) | 20.57 (10.489)
  Week 60: number analyzed (Participants) | 363 | 331
  Week 60 | 21.39 (10.139) | 20.36 (10.250)
  Week 72: number analyzed (Participants) | 339 | 304
  Week 72 | 22.56 (11.326) | 21.58 (11.225)
  Week 84: number analyzed (Participants) | 306 | 276
  Week 84 | 22.29 (9.967) | 22.30 (10.728)
  Week 96: number analyzed (Participants) | 236 | 210
  Week 96 | 22.63 (10.563) | 21.83 (10.463)
  Week 108: number analyzed (Participants) | 191 | 166
  Week 108 | 22.97 (10.305) | 22.17 (11.535)
  Week 120: number analyzed (Participants) | 148 | 132
  Week 120 | 24.45 (11.315) | 22.55 (12.332)
  Week 132: number analyzed (Participants) | 114 | 91
  Week 132 | 25.50 (11.083) | 22.33 (11.377)
  Week 144: number analyzed (Participants) | 77 | 70
  Week 144 | 25.02 (10.830) | 21.06 (9.960)
  Week 156: number analyzed (Participants) | 51 | 47
  Week 156 | 27.30 (14.396) | 21.46 (10.506)
  Week 168: number analyzed (Participants) | 35 | 24
  Week 168 | 28.87 (12.654) | 23.91 (11.704)
  Week 180: number analyzed (Participants) | 15 | 13
  Week 180 | 33.63 (15.515) | 25.72 (8.827)
  Early Term/ Discontinuation: number analyzed (Participants) | 98 | 115
  Early Term/ Discontinuation | 22.18 (13.112) | 21.32 (10.752)
  Final Visit: number analyzed (Participants) | 231 | 208
  Final Visit | 24.62 (11.311) | 24.03 (11.099)

7. Secondary Outcome: Vitamin E Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 427.067 Days), Final Visit (Mean: 908.715 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
ug/mL
  Baseline: number analyzed (Participants) | 498 | 485
  Baseline | 16.55 (6.204) | 16.29 (6.188)
  Week 12: number analyzed (Participants) | 461 | 456
  Week 12 | 16.59 (6.152) | 16.94 (6.756)
  Week 24: number analyzed (Participants) | 438 | 415
  Week 24 | 16.87 (6.146) | 16.82 (6.275)
  Week 36: number analyzed (Participants) | 411 | 397
  Week 36 | 17.32 (7.280) | 16.82 (6.046)
  Week 48: number analyzed (Participants) | 388 | 371
  Week 48 | 17.12 (6.653) | 16.95 (6.204)
  Week 60: number analyzed (Participants) | 362 | 332
  Week 60 | 16.60 (5.787) | 17.14 (6.267)
  Week 72: number analyzed (Participants) | 338 | 303
  Week 72 | 16.79 (6.188) | 17.10 (6.242)
  Week 84: number analyzed (Participants) | 306 | 274
  Week 84 | 17.13 (6.978) | 16.82 (5.847)
  Week 96: number analyzed (Participants) | 236 | 210
  Week 96 | 17.42 (6.987) | 17.21 (6.007)
  Week 108: number analyzed (Participants) | 190 | 167
  Week 108 | 17.27 (6.403) | 17.03 (5.986)
  Week 120: number analyzed (Participants) | 147 | 131
  Week 120 | 16.95 (5.217) | 16.79 (5.870)
  Week 132: number analyzed (Participants) | 114 | 92
  Week 132 | 16.81 (5.533) | 16.42 (6.081)
  Week 144: number analyzed (Participants) | 78 | 70
  Week 144 | 17.11 (6.970) | 17.06 (6.607)
  Week 156: number analyzed (Participants) | 51 | 48
  Week 156 | 16.64 (6.016) | 16.70 (6.491)
  Week 168: number analyzed (Participants) | 35 | 24
  Week 168 | 16.64 (6.435) | 18.02 (6.865)
  Week 180: number analyzed (Participants) | 15 | 13
  Week 180 | 15.57 (4.474) | 17.58 (5.239)
  Early Term/ Discontinuation: number analyzed (Participants) | 98 | 112
  Early Term/ Discontinuation | 16.32 (5.047) | 16.25 (6.334)
  Final Visit: number analyzed (Participants) | 230 | 208
  Final Visit | 15.60 (5.731) | 15.92 (6.211)

8. Secondary Outcome: Vitamin K Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 432.942 Days), Final Visit (Mean: 910.448 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
ng/mL
  Baseline: number analyzed (Participants) | 435 | 436
  Baseline | 0.663 (0.6138) | 0.628 (0.6023)
  Week 12: number analyzed (Participants) | 411 | 407
  Week 12 | 0.651 (0.6296) | 0.653 (0.6060)
  Week 24: number analyzed (Participants) | 391 | 376
  Week 24 | 0.655 (0.5999) | 0.658 (0.6364)
  Week 36: number analyzed (Participants) | 361 | 355
  Week 36 | 0.730 (0.6616) | 0.640 (0.6120)
  Week 48: number analyzed (Participants) | 356 | 336
  Week 48 | 0.626 (0.5746) | 0.649 (0.6211)
  Week 60: number analyzed (Participants) | 334 | 305
  Week 60 | 0.695 (0.6458) | 0.732 (0.6640)
  Week 72: number analyzed (Participants) | 310 | 274
  Week 72 | 0.703 (0.6295) | 0.703 (0.6668)
  Week 84: number analyzed (Participants) | 281 | 260
  Week 84 | 0.775 (0.7309) | 0.717 (0.6631)
  Week 96: number analyzed (Participants) | 221 | 196
  Week 96 | 0.723 (0.6386) | 0.682 (0.6382)
  Week 108: number analyzed (Participants) | 178 | 162
  Week 108 | 0.801 (0.7190) | 0.737 (0.7428)
  Week 120: number analyzed (Participants) | 136 | 124
  Week 120 | 0.688 (0.7177) | 0.717 (0.6918)
  Week 132: number analyzed (Participants) | 107 | 86
  Week 132 | 0.782 (0.7253) | 0.650 (0.6832)
  Week 144: number analyzed (Participants) | 76 | 66
  Week 144 | 0.661 (0.6658) | 0.662 (0.5824)
  Week 156: number analyzed (Participants) | 49 | 47
  Week 156 | 0.685 (0.6300) | 0.724 (0.6570)
  Week 168: number analyzed (Participants) | 35 | 24
  Week 168 | 0.822 (0.7662) | 0.862 (0.7611)
  Week 180: number analyzed (Participants) | 14 | 13
  Week 180 | 0.879 (0.8268) | 1.020 (1.0008)
  Early Term / Discontinuation: number analyzed (Participants) | 91 | 100
  Early Term / Discontinuation | 0.761 (0.6920) | 0.679 (0.6541)
  Final Visit: number analyzed (Participants) | 218 | 197
  Final Visit | 0.843 (0.7197) | 0.814 (0.6982)

9. Secondary Outcome: Serum Folate Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 420.569 Days), Final Visit (Mean: 909.848 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 505
ng/mL
  Baseline: number analyzed (Participants) | 489 | 487
  Baseline | 15.51 (28.300) | 18.87 (37.577)
  Week 12: number analyzed (Participants) | 458 | 450
  Week 12 | 13.46 (23.247) | 18.57 (38.500)
  Week 24: number analyzed (Participants) | 433 | 416
  Week 24 | 13.79 (28.539) | 17.44 (39.950)
  Week 36: number analyzed (Participants) | 408 | 391
  Week 36 | 13.35 (24.059) | 16.61 (34.428)
  Week 48: number analyzed (Participants) | 382 | 364
  Week 48 | 13.84 (24.193) | 18.16 (40.329)
  Week 60: number analyzed (Participants) | 355 | 327
  Week 60 | 13.25 (20.655) | 17.57 (40.427)
  Week 72: number analyzed (Participants) | 330 | 293
  Week 72 | 12.78 (21.370) | 17.76 (38.679)
  Week 84: number analyzed (Participants) | 296 | 270
  Week 84 | 12.67 (19.767) | 14.34 (26.514)
  Week 96: number analyzed (Participants) | 231 | 207
  Week 96 | 13.27 (18.484) | 17.20 (37.621)
  Week 108: number analyzed (Participants) | 188 | 163
  Week 108 | 12.76 (18.758) | 17.10 (42.133)
  Week 120: number analyzed (Participants) | 147 | 131
  Week 120 | 12.34 (13.152) | 18.93 (46.884)
  Week 132: number analyzed (Participants) | 113 | 90
  Week 132 | 12.13 (12.813) | 14.08 (36.549)
  Week 144: number analyzed (Participants) | 78 | 70
  Week 144 | 14.26 (31.355) | 9.93 (9.423)
  Week 156: number analyzed (Participants) | 51 | 46
  Week 156 | 12.12 (12.259) | 10.04 (10.910)
  Week 168: number analyzed (Participants) | 35 | 24
  Week 168 | 13.90 (16.225) | 17.62 (31.941)
  Week 180: number analyzed (Participants) | 15 | 13
  Week 180 | 16.63 (17.402) | 13.45 (14.884)
  Early Term/ Discontinuation: number analyzed (Participants) | 93 | 111
  Early Term/ Discontinuation | 12.28 (18.101) | 23.21 (35.035)
  Final Visit: number analyzed (Participants) | 230 | 204
  Final Visit | 13.62 (24.370) | 18.36 (42.611)

ADVERSE EVENTS:
Description: The AE analysis is based on the Safety Population. The Safety Population included all patients who were randomized and received at least 1 dose of study drug. The start number of Participant Flow included all patients who were randomized.
Arm/Group | AST-120 | Placebo
Serious Adverse Events (participants affected / at risk) | 156/507 | 178/505
Other Adverse Events (participants affected / at risk) | 393/507 | 377/505
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AST-120 (N=507) | Placebo (N=505)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 8 | 6
Angina pectoris (Cardiac disorders) | 2 | 5
Angina unstable (Cardiac disorders) | 5 | 4
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 1
Atrial flutter (Cardiac disorders) | 2 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 4
Cardiac arrest (Cardiac disorders) | 3 | 3
Cardiac failure (Cardiac disorders) | 4 | 4
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 11
Cardiogenic shock (Cardiac disorders) | 0 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiomyopathy alcoholic (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 3
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1
Myxoedema (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 4
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Device difficult to use (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Device lead damage (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Necrobiosis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 2
Oedema (General disorders) | 1 | 0
Oedema due to renal disease (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Sudden cardiac death (General disorders) | 2 | 0
Sudden death (General disorders) | 0 | 4
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 4
Bronchitis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 4 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diabetic gangrene (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2
Escherichia urinary tract infection (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 2
Myringitis bullous (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 4
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 3
Septic shock (Infections and infestations) | 2 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 6
Urosepsis (Infections and infestations) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Chest X-ray abnormal (Investigations) | 1 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 3
Diabetic foot (Metabolism and nutrition disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 1
Cerebral circulatory failure (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 7 | 5
Convulsion (Nervous system disorders) | 1 | 1
Encephalomyelitis (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 2
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Radiculitis lumbosacral (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Azotaemia (Renal and urinary disorders) | 5 | 4
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 2
Renal failure acute (Renal and urinary disorders) | 14 | 13
Renal failure chronic (Renal and urinary disorders) | 34 | 47
Renal impairment (Renal and urinary disorders) | 0 | 4
Urinary retention (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 9 | 11
Catheter placement (Surgical and medical procedures) | 0 | 1
Central venous catheterisation (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Dialysis device insertion (Surgical and medical procedures) | 0 | 1
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 2 | 4
Obesity surgery (Surgical and medical procedures) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 6 | 8
Hypertensive crisis (Vascular disorders) | 3 | 4
Hypertensive emergency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 2
Ischaemia (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AST-120 (N=507) | Placebo (N=505)
Anaemia (Blood and lymphatic system disorders) | 75 | 83
Angina pectoris (Cardiac disorders) | 1 | 7
Vertigo (Ear and labyrinth disorders) | 2 | 6
Hyperparathyroidism (Endocrine disorders) | 7 | 4
Hyperparathyroidism secondary (Endocrine disorders) | 9 | 8
Cataract (Eye disorders) | 12 | 6
Eye haemorrhage (Eye disorders) | 7 | 0
Abdominal discomfort (Gastrointestinal disorders) | 9 | 0
Abdominal distension (Gastrointestinal disorders) | 16 | 16
Abdominal pain (Gastrointestinal disorders) | 18 | 19
Abdominal pain upper (Gastrointestinal disorders) | 14 | 13
Constipation (Gastrointestinal disorders) | 55 | 38
Diarrhoea (Gastrointestinal disorders) | 42 | 41
Dyspepsia (Gastrointestinal disorders) | 16 | 21
Faeces discoloured (Gastrointestinal disorders) | 4 | 11
Flatulence (Gastrointestinal disorders) | 12 | 15
Gastritis (Gastrointestinal disorders) | 20 | 22
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 2
Nausea (Gastrointestinal disorders) | 45 | 45
Vomiting (Gastrointestinal disorders) | 28 | 36
Asthenia (General disorders) | 14 | 20
Chest pain (General disorders) | 7 | 6
Chills (General disorders) | 6 | 1
Fatigue (General disorders) | 22 | 14
Oedema (General disorders) | 13 | 13
Oedema peripheral (General disorders) | 46 | 57
Pyrexia (General disorders) | 8 | 9
Bronchitis (Infections and infestations) | 14 | 19
Cellulitis (Infections and infestations) | 7 | 5
Cystitis (Infections and infestations) | 6 | 4
Gastroenteritis (Infections and infestations) | 9 | 6
Herpes zoster (Infections and infestations) | 7 | 3
Influenza (Infections and infestations) | 26 | 21
Nasopharyngitis (Infections and infestations) | 21 | 14
Pharyngitis (Infections and infestations) | 11 | 8
Pneumonia (Infections and infestations) | 5 | 6
Respiratory tract infection (Infections and infestations) | 9 | 9
Respiratory tract infection viral (Infections and infestations) | 4 | 6
Sinusitis (Infections and infestations) | 14 | 5
Upper respiratory tract infection (Infections and infestations) | 25 | 19
Urinary tract infection (Infections and infestations) | 28 | 33
Contusion (Injury, poisoning and procedural complications) | 8 | 2
Fall (Injury, poisoning and procedural complications) | 6 | 5
Blood bicarbonate decreased (Investigations) | 7 | 3
Blood creatine phosphokinase increased (Investigations) | 12 | 9
Blood pressure increased (Investigations) | 10 | 9
Weight increased (Investigations) | 6 | 3
Acidosis (Metabolism and nutrition disorders) | 4 | 7
Decreased appetite (Metabolism and nutrition disorders) | 15 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 6 | 4
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 7
Gout (Metabolism and nutrition disorders) | 24 | 19
Hypercalcaemia (Metabolism and nutrition disorders) | 7 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 14
Hyperkalaemia (Metabolism and nutrition disorders) | 43 | 35
Hyperphosphataemia (Metabolism and nutrition disorders) | 22 | 17
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 12 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6
Metabolic acidosis (Metabolism and nutrition disorders) | 17 | 14
Vitamin D deficiency (Metabolism and nutrition disorders) | 15 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 | 27
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 16
Dizziness (Nervous system disorders) | 16 | 15
Headache (Nervous system disorders) | 17 | 21
Hypoaesthesia (Nervous system disorders) | 7 | 0
Anxiety (Psychiatric disorders) | 9 | 5
Depression (Psychiatric disorders) | 9 | 12
Insomnia (Psychiatric disorders) | 14 | 13
Haematuria (Renal and urinary disorders) | 1 | 6
Proteinuria (Renal and urinary disorders) | 6 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 6
Renal failure chronic (Renal and urinary disorders) | 40 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 21
Dermatitis (Skin and subcutaneous tissue disorders) | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 18
Rash (Skin and subcutaneous tissue disorders) | 9 | 12
Arteriovenous fistula operation (Surgical and medical procedures) | 16 | 22
Hypertension (Vascular disorders) | 54 | 49
Hypertensive crisis (Vascular disorders) | 7 | 2
Hypotension (Vascular disorders) | 15 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other